CLINICAL TRIAL: NCT03985670
Title: Neoadjuvant Teripalimab Plus Chemotherapy in Local Advanced Esophageal Squamous Cancer
Brief Title: Teripalimab Plus Chemotherapy in Local Advanced Esophageal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HenanCH immunotherapy001
Record Dates: First submitted 2019-06-10; First posted 2019-06-14 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-06

CONDITIONS: Squamous Cell Carcinoma; Esophageal Cancer; Perioperative Period
MeSH Terms: conditions — Carcinoma, Squamous Cell; Esophageal Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Intervention Model Description: patients with local advanced esophageal squamous cell carcinoma receive two cycle of neoadjuvant chemotherapy and PD-1 antibody in the same day or chemotherapy followed by PD-1 antibody, and then surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment group (Experimental): teripalimab 240mg d1 paclitaxel 150-175mg/m2 d1 cisplatin 70-75mg/m2 d1
  Interventions: Drug: teripalimab plus chemotherapy
- chemotherapy followed by immunotherapy (Active Comparator): paclitaxel 150-175mg/m2 d1 cisplatin 70-75mg/m2 d1 teripalimab 240mg d3
  Interventions: Drug: chemotherapy plus teripalimab

INTERVENTIONS:
Drug: teripalimab plus chemotherapy — teripalimab 240mg d1 paclitaxel 150mg/m2 d1 cisplatin 70mg/m2 d1
  Other Names: teripalimab and chemotherapy given on the same day
  Arms: treatment group
Drug: chemotherapy plus teripalimab — paclitaxel 150mg/m2 d1 cisplatin 70mg/m2 d1 teripalimab 240mg d3
  Other Names: chemotherapy followed by teripalimab
  Arms: chemotherapy followed by immunotherapy

SUMMARY:
The prognosis of locally advanced esophageal squamous cell carcinoma is poor,the role of chemotherapy as neoadjuvant therapy in locally advanced esophageal cancer has been established, which can convert some unresectable esophageal cancer into resectable esophageal cancer.PD-1 antibody has been shown to improve the pathological complete response rate in NSCLC, however, the data in neoadjuvant of esophageal squamous carcinoma is relatively rare. This study was designed to know the value of PD-1 antibody in neoadjuvant therapy of esophageal cancer.

DETAILED DESCRIPTION:
The prognosis of locally advanced esophageal squamous cell carcinoma is poor, the 5-year survival rate is less than 50%. It is necessary to conduct studies in these patients to reduce the rate of postoperative recurrence and prolong the disease-free survival. The role of chemotherapy as neoadjuvant therapy in locally advanced esophageal cancer has been established, which can convert some unresectable esophageal cancer into resectable esophageal cancer. The PD-1 antibody, teripalimab, is an immunological checkpoint inhibitor that has shown clinical efficacy in advanced esophageal cancer, but there has been relatively few data on neoadjuvant therapy. This study was designed to comprehend the pathological complete response rate, disease-free survival, and safety of neoadjuvant therapy with chemotherapy plus teriprilin patients with locally advanced esophageal squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Thoracic esophageal squamous cell carcinoma diagnosed by pathology
* no distant metastasis, the diseases could be resected or potentially resectable assessed by thoracic oncologist
* ECOG score 0-1
* clinical stage is stage II, III, and IVa according to AJCC 8.0
* expected lifespan > 3 months
* enough organ function
* normal blood pressure, for patients with hypertension, the blood pressure should be controlled in normal level by antihypertension
* the fasting blood sugar should be ≤ 8mmol / L for diabetic patients
* no other serious diseases (such as autoimmune diseases, immunodeficiencies, organ transplants) that conflict with this study
* no history of other malignant tumors
* women of childbearing period must be tested negative for blood pregnancy within 7 days, and subjects of childbearing age must use appropriate contraceptive measures during the trial period and within 6 months after the trial;
* The patient agrees to participate in the clinical study and sign the Informed Consent Form.

Exclusion Criteria:

* suffering from serious infectious diseases within 4 weeks before enrollment;
* patients with bronchial asthma requires intermittent use of bronchodilators or medical interventions;
* usage of immunosuppressants before the enrollment, the amount of immunosuppressant used ≥10mg / day oral prednisone for more than 2 weeks
* clinically significant cardiovascular and cerebrovascular diseases, including but not limited to severe acute myocardial infarction, unstable or severe angina, coronary artery bypass surgery, congestive heart failure, and room requiring medical intervention within the first 6 months of enrollment arrhythmia, left ventricular ejection fraction <50%
* severe allergies
* severe mental disorder
* abnormal blood coagulation function (PT>16s, APTT>53s, TT>21s, Fib<1.5g/L), bleeding tendency or receiving thrombolysis or anticoagulant therapy
* previous or current pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, severe lung damage, etc
* other situations evaluated by investigators not meet the enrollment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-07-10 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate | two months
  the proportion of patients got pathological complete response rate

SECONDARY OUTCOMES:
occurrence rate of adverse events | three month
  the occurrence of adverse events
disease-free survival rate | three years
  the proportion of patients without relapse

CONTACTS AND LOCATIONS:
Overall Officials: Jing Ding, Master, Principal Investigator — Henan Cancer Hospital
Locations (1):
- Affiliated Cancer Hospital of Zhengzhou University & Henan Cancer Hospital, Zhengzhou, Henan, China

REFERENCES:
- [Derived] Xing W, Zhao L, Zheng Y, Liu B, Liu X, Li T, Zhang Y, Ma B, Yang Y, Shang Y, Fu X, Liang G, Yuan D, Qu J, Chai X, Zhang H, Wang Z, Lin H, Liu L, Ren X, Zhang J, Gao Q. The Sequence of Chemotherapy and Toripalimab Might Influence the Efficacy of Neoadjuvant Chemoimmunotherapy in Locally Advanced Esophageal Squamous Cell Cancer-A Phase II Study. Front Immunol. 2021 Dec 6;12:772450. doi: 10.3389/fimmu.2021.772450. eCollection 2021. PMID 34938292
- [Derived] Xing W, Zhao L, Fu X, Liang G, Zhang Y, Yuan D, Li Z, Gao Q, Zheng Y; written on Henan Cancer Hospital Thoracic Oncology Group (HCHTOG). A phase II, single-centre trial of neoadjuvant toripalimab plus chemotherapy in locally advanced esophageal squamous cell carcinoma. J Thorac Dis. 2020 Nov;12(11):6861-6867. doi: 10.21037/jtd-20-2198. PMID 33282388